CLINICAL TRIAL: NCT05278923
Title: The Impact of Soiled Airway Management on CPR Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20180503R
Record Dates: First submitted 2022-02-17; First posted 2022-03-14 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-02

CONDITIONS: Airway Aspiration; Cardiopulmonary Arrest
Keywords: resuscitation, Airway decontamination, suction assisted
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Two scenarios were simulated. CPR and ETI in an airway with regurgitation (oropharyngeal regurgitation scenario) and CPR and ETI in an airway without regurgitation (clean airway scenario). All EMT-Ps were assigned to participate initially in one of the scenarios. After all EMT-Ps had finished the first scenario, they switched to the other.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clean airway (No Intervention): CPR and endotracheal intubation in an airway without regurgitation
- regurgitation airway (Experimental): CPR and endotracheal intubation in an airway with regurgitation
  Interventions: Device: SALAD simulation device

INTERVENTIONS:
Device: SALAD simulation device — An airway CPR manikin was modified to simulate regurgitation during CPR . A manual pump was fixed on the bottom of the torso to simulate the stomach. A clear vinyl tube was connected the manikin's oesophagus and the outflow port of the pump. A water container outside the manikin was filled with simulated gastric content and connected to the inflow port of the pump through another vinyl tube. The manikin's left main bronchus was occluded using a red cap provided by the manufacturer. The lung was simulated by an anaesthesia breathing bag placed outside the manikin and connected to the manikin's right main bronchus via a breathing circuit. A compression pad was attached to the bottom of the manikin's compression plate. During chest compression, the compression pad squeezed the pump to regurgitate gastric contents into the oropharynx
  Arms: regurgitation airway

SUMMARY:
Regurgitation is an adverse event common during cardiopulmonary resuscitation (CPR) and occurs in 20%-32% of patients experiencing out-of-hospital cardiac arrest (OHCA). It can impair ventilation, induce aspiration, and decrease survival to hospital discharge. Gastric fluid in the airway obscures the laryngeal view, thereby considerably decreasing the first-pass success of endotracheal intubation (ETI) by paramedics.

A human cadaver study reported that ETI outperforms other airway management devices, such as the i-gel, laryngeal mask, and laryngeal tube, in preventing aspiration when regurgitation occurs during CPR. However, ETI is also associated with multiple and prolonged CPR pauses.Compared with the use of supraglottic airway (SGA) devices, ETI results in more hands-off time during CPR. Recent randomised clinical trials have revealed that airway management with an SGA device provides superior outcomes to those of ETI in patients with OHCA. However, ETI remains the preferred management strategy for an airway affected by regurgitation in patients with OHCA.

Current guidelines focus on the quality of CPR because it is a key determinant of survival in patients with OHCA. However, evidence regarding the impact of regurgitation during ETI on CPR quality is limited. This manikin simulation study assessed CPR quality during ETI in airways with and without regurgitation.

DETAILED DESCRIPTION:
This is a prospective compare study. 54 EMT-Ps, are involved to evaluate the impact of airway management on CPR quality.

The Study uses SALAD training tool for training. The SALAD training tool include Nasco Intubation CPR manikin, which could vomit by pumping liquid into distal esophagus, and HQCPR feedback machine. Two scenarios were simulated. CPR and ETI in an airway with regurgitation (oropharyngeal regurgitation scenario) and CPR and ETI in an airway without regurgitation (clean airway scenario). All EMT-Ps were randomly assigned to participate initially in one of the scenarios. After all EMT-Ps had finished the first scenario, they switched to the other. Three EMT-Ps formed a resuscitation team and played one of the following roles: airway manager, first compressor, or second compressor. In each scenario, each EMT-P was required to take a turn playing all three roles. During each simulation, the airway manager performed BVM ventilation, and the first and second compressors alternately provided chest compression for every five cycles of CPR, with a compression-to-ventilation ratio of 30:2 .

After the first five cycles of CPR, the airway manager was asked to perform intubation during the ongoing chest compression to minimise intubation-associated interruption of chest compression. If necessary, the airway manager could request a pause of the ongoing chest compression. If intubation was not successful, the airway manager performed BVM ventilation twice and then reattempt intubation. After intubation, the airway manager used the BVM to check the lung distention to confirm successful intubation. Each simulation was ended after successful or failed intubation. Failed intubation was defined as either oesophageal intubation or three unsuccessful attempts.

The primary outcomes was chest compression fraction (CCF). The secondary outcomes was the intubation success rate. Chest compression depth, chest compression rate, and longest interruption time, and intubation time were also recorded.

Each CPR-intubation sequence comprised two segments: a compression segment and a hands-off segment. CCF was defined as the proportion of time spent on chest compression in each CPR-intubation sequence. The longest interruption time was defined as the longest hands-off duration in each sequence. An intubation attempt was defined as the insertion of the laryngoscope blade into the mouth and its subsequent withdrawal from the mouth. Intubation time was defined as the period between the start and the end of an intubation attempt. The time spent checking the endotracheal tube position by manual ventilation through the endotracheal tube was not included in the CPR-intubation sequence.

Two video cameras were setup to record the entire simulation process. Two observers reviewed the video records independently to identify the start and end of each CPR-intubation sequence, any intubation attempts, and the hands-off and compression segments of each sequence. Disagreements were resolved by reaching mutual consensus. The HQCPR application on an Android device recorded chest compression depth, rate, and interruptions (defined as no chest compression [hands off] for >1 s). The data from both the video recording and the HQCPR application were used in subsequent analysis.Continuous data are presented as medians with interquartile ranges, and categorical data are presented as frequency counts and percentages. The continuous data were compared using the Wilcoxon rank sum test in the first CPR-intubation sequence and the Mann-Whitney U test in the second and third sequences. The McNemar test was used to compare the intubation success rate in the first sequence, and Pearson's chi-square test was used for the second and third sequences. The continuous data from all three CPR-intubation sequences were compared using the Kruskal-Wallis test. Post hoc analysis was performed using Conover's test.

The association of CPR quality metrics with successful intubation was evaluated using a Cox proportional hazards regression model. The results of multivariate analyses are presented as hazard ratios (HRs) with corresponding 95% confidence intervals (CIs). A two-tailed P <0.05 indicates statistical significance. MedCalc Statistical Software version 19.2. (MedCalc Software, Ostend, Belgium) was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* emergency medical technician-paramedics experienced in advanced airway management and CPR

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
chest compression fraction | 3 hours
  the proportion of time spent performing chest compressions during arrest

SECONDARY OUTCOMES:
intubation success rate | 3 hours
  the rate of successful intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Shinkong Wu-Ho-Su memorial hospital, Taipei, Shih-Lin, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simons RW, Rea TD, Becker LJ, Eisenberg MS. The incidence and significance of emesis associated with out-of-hospital cardiac arrest. Resuscitation. 2007 Sep;74(3):427-31. doi: 10.1016/j.resuscitation.2007.01.038. Epub 2007 Apr 11. PMID 17433526
- [Background] Virkkunen I, Kujala S, Ryynanen S, Vuori A, Pettila V, Yli-Hankala A, Silfvast T. Bystander mouth-to-mouth ventilation and regurgitation during cardiopulmonary resuscitation. J Intern Med. 2006 Jul;260(1):39-42. doi: 10.1111/j.1365-2796.2006.01664.x. PMID 16789977
- [Background] Virkkunen I, Ryynanen S, Kujala S, Vuori A, Piilonen A, Kaaria JP, Kahara V, Pettila V, Yli-Hankala A, Silfvast T. Incidence of regurgitation and pulmonary aspiration of gastric contents in survivors from out-of-hospital cardiac arrest. Acta Anaesthesiol Scand. 2007 Feb;51(2):202-5. doi: 10.1111/j.1399-6576.2006.01229.x. PMID 17261147
- [Background] Prekker ME, Kwok H, Shin J, Carlbom D, Grabinsky A, Rea TD. The process of prehospital airway management: challenges and solutions during paramedic endotracheal intubation. Crit Care Med. 2014 Jun;42(6):1372-8. doi: 10.1097/CCM.0000000000000213. PMID 24589641
- [Background] Piegeler T, Roessler B, Goliasch G, Fischer H, Schlaepfer M, Lang S, Ruetzler K. Evaluation of six different airway devices regarding regurgitation and pulmonary aspiration during cardio-pulmonary resuscitation (CPR) - A human cadaver pilot study. Resuscitation. 2016 May;102:70-4. doi: 10.1016/j.resuscitation.2016.02.017. Epub 2016 Feb 26. PMID 26921473
- [Background] Wang HE, Simeone SJ, Weaver MD, Callaway CW. Interruptions in cardiopulmonary resuscitation from paramedic endotracheal intubation. Ann Emerg Med. 2009 Nov;54(5):645-652.e1. doi: 10.1016/j.annemergmed.2009.05.024. Epub 2009 Jul 2. PMID 19573949
- [Background] Kurz MC, Prince DK, Christenson J, Carlson J, Stub D, Cheskes S, Lin S, Aziz M, Austin M, Vaillancourt C, Colvin J, Wang HE; ROC Investigators. Association of advanced airway device with chest compression fraction during out-of-hospital cardiopulmonary arrest. Resuscitation. 2016 Jan;98:35-40. doi: 10.1016/j.resuscitation.2015.10.011. Epub 2015 Oct 28. PMID 26520783
- [Background] Ruetzler K, Gruber C, Nabecker S, Wohlfarth P, Priemayr A, Frass M, Kimberger O, Sessler DI, Roessler B. Hands-off time during insertion of six airway devices during cardiopulmonary resuscitation: a randomised manikin trial. Resuscitation. 2011 Aug;82(8):1060-3. doi: 10.1016/j.resuscitation.2011.03.027. Epub 2011 Apr 6. PMID 21514986
- [Background] Wang HE, Schmicker RH, Daya MR, Stephens SW, Idris AH, Carlson JN, Colella MR, Herren H, Hansen M, Richmond NJ, Puyana JCJ, Aufderheide TP, Gray RE, Gray PC, Verkest M, Owens PC, Brienza AM, Sternig KJ, May SJ, Sopko GR, Weisfeldt ML, Nichol G. Effect of a Strategy of Initial Laryngeal Tube Insertion vs Endotracheal Intubation on 72-Hour Survival in Adults With Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2018 Aug 28;320(8):769-778. doi: 10.1001/jama.2018.7044. PMID 30167699
- [Background] Voss S, Rhys M, Coates D, Greenwood R, Nolan JP, Thomas M, Benger J. How do paramedics manage the airway during out of hospital cardiac arrest? Resuscitation. 2014 Dec;85(12):1662-6. doi: 10.1016/j.resuscitation.2014.09.008. Epub 2014 Sep 26. PMID 25260723
- [Background] Nolan JP, Maconochie I, Soar J, Olasveengen TM, Greif R, Wyckoff MH, Singletary EM, Aickin R, Berg KM, Mancini ME, Bhanji F, Wyllie J, Zideman D, Neumar RW, Perkins GD, Castren M, Morley PT, Montgomery WH, Nadkarni VM, Billi JE, Merchant RM, de Caen A, Escalante-Kanashiro R, Kloeck D, Wang TL, Hazinski MF. Executive Summary: 2020 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2020 Oct 20;142(16_suppl_1):S2-S27. doi: 10.1161/CIR.0000000000000890. Epub 2020 Oct 21. No abstract available. PMID 33084397
- [Background] Meaney PA, Bobrow BJ, Mancini ME, Christenson J, de Caen AR, Bhanji F, Abella BS, Kleinman ME, Edelson DP, Berg RA, Aufderheide TP, Menon V, Leary M; CPR Quality Summit Investigators, the American Heart Association Emergency Cardiovascular Care Committee, and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Cardiopulmonary resuscitation quality: [corrected] improving cardiac resuscitation outcomes both inside and outside the hospital: a consensus statement from the American Heart Association. Circulation. 2013 Jul 23;128(4):417-35. doi: 10.1161/CIR.0b013e31829d8654. Epub 2013 Jun 25. PMID 23801105
- [Background] DuCanto J, Serrano KD, Thompson RJ. Novel Airway Training Tool that Simulates Vomiting: Suction-Assisted Laryngoscopy Assisted Decontamination (SALAD) System. West J Emerg Med. 2017 Jan;18(1):117-120. doi: 10.5811/westjem.2016.9.30891. Epub 2016 Nov 8. PMID 28116021
- [Background] Root CW, Mitchell OJL, Brown R, Evers CB, Boyle J, Griffin C, West FM, Gomm E, Miles E, McGuire B, Swaminathan A, St George J, Horowitz JM, DuCanto J. Suction Assisted Laryngoscopy and Airway Decontamination (SALAD): A technique for improved emergency airway management. Resusc Plus. 2020 May 21;1-2:100005. doi: 10.1016/j.resplu.2020.100005. eCollection 2020 Mar-Jun. PMID 34223292
- [Background] Christenson J, Andrusiek D, Everson-Stewart S, Kudenchuk P, Hostler D, Powell J, Callaway CW, Bishop D, Vaillancourt C, Davis D, Aufderheide TP, Idris A, Stouffer JA, Stiell I, Berg R; Resuscitation Outcomes Consortium Investigators. Chest compression fraction determines survival in patients with out-of-hospital ventricular fibrillation. Circulation. 2009 Sep 29;120(13):1241-7. doi: 10.1161/CIRCULATIONAHA.109.852202. Epub 2009 Sep 14. PMID 19752324
- [Background] Rea T, Olsufka M, Yin L, Maynard C, Cobb L. The relationship between chest compression fraction and outcome from ventricular fibrillation arrests in prolonged resuscitations. Resuscitation. 2014 Jul;85(7):879-84. doi: 10.1016/j.resuscitation.2014.02.026. Epub 2014 Mar 4. PMID 24607869
- [Background] Vaillancourt C, Petersen A, Meier EN, Christenson J, Menegazzi JJ, Aufderheide TP, Nichol G, Berg R, Callaway CW, Idris AH, Davis D, Fowler R, Egan D, Andrusiek D, Buick JE, Bishop TJ, Colella MR, Sahni R, Stiell IG, Cheskes S; Resuscitation Outcomes Consortium Investigators.. The impact of increased chest compression fraction on survival for out-of-hospital cardiac arrest patients with a non-shockable initial rhythm. Resuscitation. 2020 Sep;154:93-100. doi: 10.1016/j.resuscitation.2020.06.016. Epub 2020 Jun 20. PMID 32574654
- [Background] Vadeboncoeur T, Stolz U, Panchal A, Silver A, Venuti M, Tobin J, Smith G, Nunez M, Karamooz M, Spaite D, Bobrow B. Chest compression depth and survival in out-of-hospital cardiac arrest. Resuscitation. 2014 Feb;85(2):182-8. doi: 10.1016/j.resuscitation.2013.10.002. Epub 2013 Oct 12. PMID 24125742
- [Background] Kleinman ME, Brennan EE, Goldberger ZD, Swor RA, Terry M, Bobrow BJ, Gazmuri RJ, Travers AH, Rea T. Part 5: Adult Basic Life Support and Cardiopulmonary Resuscitation Quality: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S414-35. doi: 10.1161/CIR.0000000000000259. No abstract available. PMID 26472993
- [Background] Michalek P, Donaldson W, Vobrubova E, Hakl M. Complications Associated with the Use of Supraglottic Airway Devices in Perioperative Medicine. Biomed Res Int. 2015;2015:746560. doi: 10.1155/2015/746560. Epub 2015 Dec 13. PMID 26783527
- [Background] Benger JR, Kirby K, Black S, Brett SJ, Clout M, Lazaroo MJ, Nolan JP, Reeves BC, Robinson M, Scott LJ, Smartt H, South A, Stokes EA, Taylor J, Thomas M, Voss S, Wordsworth S, Rogers CA. Effect of a Strategy of a Supraglottic Airway Device vs Tracheal Intubation During Out-of-Hospital Cardiac Arrest on Functional Outcome: The AIRWAYS-2 Randomized Clinical Trial. JAMA. 2018 Aug 28;320(8):779-791. doi: 10.1001/jama.2018.11597. PMID 30167701
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Fevang E, Haaland K, Roislien J, Bjorshol CA. Semiprone position is superior to supine position for paediatric endotracheal intubation during massive regurgitation, a randomized crossover simulation trial. BMC Anesthesiol. 2018 Jan 18;18(1):10. doi: 10.1186/s12871-018-0474-z. PMID 29347980
- [Background] Sorour K, Donovan L. Intentional esophageal intubation to improve visualization during emergent endotracheal intubation in the context of massive vomiting: a case report. J Clin Anesth. 2015 Mar;27(2):168-9. doi: 10.1016/j.jclinane.2014.07.004. Epub 2015 Jan 7. PMID 25577031
- [Background] Kornhall DK, Almqvist S, Dolven T, Ytrebo LM. Intentional oesophageal intubation for managing regurgitation during endotracheal intubation. Anaesth Intensive Care. 2015 May;43(3):412-4. No abstract available. PMID 25943615
- [Background] Lin LW, Huang CC, Ong JR, Chong CF, Wu NY, Hung SW. The suction-assisted laryngoscopy assisted decontamination technique toward successful intubation during massive vomiting simulation: A pilot before-after study. Medicine (Baltimore). 2019 Nov;98(46):e17898. doi: 10.1097/MD.0000000000017898. PMID 31725637
- [Background] Pilbery R, Teare MD. Soiled airway tracheal intubation and the effectiveness of decontamination by paramedics (SATIATED): a randomised controlled manikin study. Br Paramed J. 2019 Jun 1;4(1):14-21. doi: 10.29045/14784726.2019.06.4.1.14. PMID 33328824
- [Derived] Lin LW, DuCanto J, Hsu CY, Su YC, Huang CC, Hung SW. Compromised cardiopulmonary resuscitation quality due to regurgitation during endotracheal intubation: a randomised crossover manikin simulation study. BMC Emerg Med. 2022 Jul 9;22(1):124. doi: 10.1186/s12873-022-00662-0. PMID 35810275

DOCUMENTS (1):
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT05278923/Prot_000.pdf